CLINICAL TRIAL: NCT02418364
Title: Randomised ,Blind, Placebo Controlled in Meir Center. Study the Potential of Reflexology Treatments to Help Implant Pregnancy in Ivf Patients
Brief Title: The Effect of Reflexology Treatments on IVF Outcome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Clalit Health Services (Other); Reidman college (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0020-15
Record Dates: First submitted 2015-03-04; First posted 2015-04-16 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- placebo reflexology (Placebo Comparator): Placebo reflexology treatment
  Interventions: Other: Placebo reflexology treatment
- control group (No Intervention): Data will be taken from questionnaires
- reflexology treatment (Experimental): Reflexology treatment
  Interventions: Other: Reflexology treatment

INTERVENTIONS:
Other: Placebo reflexology treatment — Placebo reflexology treatment will be done in the same rate as the reflexology treatment itself, but will be superficial in particular,and will be directed to organs and organ systems which are not relevant to the research topic.
  Arms: placebo reflexology
Other: Reflexology treatment — Reflexology treatment will be done until the eggs implant. If the patient is not pregnant, she will start another reflexology treatment cycle. There will be minimum 4 and up to 6 reflexology treatments in every IVF cycle (maximum three IVF cycles) . Rate treatment will be two or three times a week.
  Arms: reflexology treatment

SUMMARY:
Infertility is expressed as an inability to conceive or carry a healthy pregnancy to the end. It is often said that the couple suffers from infertility if for a year they could not get a normal pregnancy. 30% of the reasons for this unsuccess are attributed to women, 30% are attributed to men, while the other 40% of cases are attributed to the combination between men and women and for unknown reasons. In women, the source of most of the problems of infertility are associated with different failures in ovulation (early ovulation, lack of ovulation or irregular ovulation). Other reasons are Blocked fallopian tubes (due to endometriosis, infection or surgery), problems in the uterus and endometrium. There is a group of women that apparently does not have the failures described above, and they have infertility that does not include pathological findings. Apparently chronic stress is a potential cause among couples who could not get pregnant (despite 6 months of focused sex) so there is a request for various techniques for reducing stress including yoga and meditation. One common option in various conditions of infertility is in vitro fertilization. This technique is also known as artificial insemination and is the most common technique used in Israel. Data from the Ministry of Health from the last years, indicate that the rate of successful pregnancies after embryo transfer is more than a third (in average), this is from an average of 20 treatment cycles.

Researches in alternative medicine are not easy to carry out. The placebo group which is usually the control group tend to be a treatment group by itself and gives effective results than a group that does not receive treatment at all. Carrying out a strict study with a good control group such as reflexology research in multiple sclerosis, has brought significant results in various statistical measures examined in this study (movement, sensory mode and urinary tract symptoms).

In the control group the calf was chosen as a place of a massage as a dummy treatment (gynecological place), which prevented contact with specific points of the feet like in patients in the treatment group. This study wishes to answer the research question: Does reflexology treatment increase the chances of pregnancy implantation in women without pathological findings that are treated with IVF. Other questions related to measures that could lead to the implant of pregnancy, are whether reflexology treatment affect the endometrial thickness, number of oocytes and embryo quality. Literature indicates the potential of reflexology treatment on ovulation induction (But requires a good control group and large sample size).

DETAILED DESCRIPTION:
The purpose of the study:

Does reflexology treatment increase the chance of pregnancy in women treated with IVF?

Research design:

To the Study will recruited women who come for IVF treatments.

Women who are fit to participate and give their consent, will be randomized to one of three treatment groups:

Group 1 - placebo reflexology

Group 2 - control group that receives no alternative treatment. Data will be taken from questionnaires

Group 3 - will be receiving a built-in protocol reflexology treatment

Reflexology treatment can begin at any stage up to the stage of the eggs implantation. If the patient is not pregnant, she will start another reflexology treatment cycle. Reflexology treatment will be minimum 4 treatments and up to six treatments for every cycle. Rate treatment will be two or three times a week. The patient can receive reflexology treatment for three cycles of IVF.

Research tools and methods

* Photo of feet before the first treatment and before final treatment
* Permanent set by 4 parameters
* Questionnaire: to be transferred at baseline and after treatment and will be in a state of double blinded. There will be no connection between the treatment protocol and questionnaires. At the end of the study, the analysis and cross checking data will form their own measurements.

  1. Quality of Life Questionnaire
  2. Questionnaire "dhak"
  3. Mind-body questionnaire
  4. Family support questionnaire

Medical tests (measurements taken any way and will be used for the study): blood tests, medical record indicating that there is no pathological findings, ultrasound, endometrial thickness, number of follicles, number of oocytes and embryo quality.

Evaluation of Participants:

80 - experimental group 80 - a control group that receives no alternative treatment 80 - a group that receives a placebo treatments

Duration of participation in the study: Six months

Treatment protocol:

The treatment strengthens the natural healing of the body, in that it strengthens the blood flow and the release of endorphins, which can reduce pain, stress relaxation and a general feeling better (wellbeing). Recently a promising theory was added, a theory called Nerve Impulse the suggests that pressure points in the foot improve neural connection to other parts of the body through the autonomic nervous system. The autonomic nervous system, regulates body systems that are under unaware control such as respiratory, heart rate and blood pressure systems which are sensitive to pressure and vibration in accordance with Physical and psychological changes, and able to control the sympathetic system and moderate the fight or flight response. Recent meta-analysis that scanned many articles pointed out that there is no unity in studies about reflexology, that there are a wide range of parameters, methods and measurements of efficacy .Therapeutic Touch are complex and it is difficult to maintain such double-blind trials.

Therefore, there is a great need for maintaining the uniformity of treatment. In the investigators' study, will be responsible coordinator of reflexology, Rachel Hoddov, to teach and train coaches participating in the study protocol the standard treatment in a way that will allow a free hand. In addition, Placebo treatment will be in superficial areas in particular, and will be directed to organs and organ systems which are not relevant to the research topic.

ELIGIBILITY:
Inclusion Criteria:

1. women age 18 To 42
2. women who receive IVF treatment
3. The number of IVF cycles - up to 7 cycles
4. Signing an informed consent form.
5. patient is required to receive at least 4 reflexology treatments until the eggs implant.

Exclusion criteria:

1. Women under 18 or over 42
2. patients who had 7 cycles of IVF

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
number of pregnant women in women treated with implantation in IVF | 6 Months
  Does reflexology treatment increase the number of pregnant women in women treated with implantation in IVF

SECONDARY OUTCOMES:
endometrial thickness | 6 months
number of oocytes | 6 months
embryo quality | 6 months
  Embryo quality measured according to the ESHRE score. Grades 1-4

REFERENCES:
- [Background] Templeton A. Infertility-epidemiology, aetiology and effective management. Health Bull (Edinb). 1995 Sep;53(5):294-8. PMID 7490200
- [Background] Ernst E. Is reflexology an effective intervention? A systematic review of randomised controlled trials. Med J Aust. 2009 Sep 7;191(5):263-6. doi: 10.5694/j.1326-5377.2009.tb02780.x. PMID 19740047
- [Background] Poole H, Glenn S, Murphy P. A randomised controlled study of reflexology for the management of chronic low back pain. Eur J Pain. 2007 Nov;11(8):878-87. doi: 10.1016/j.ejpain.2007.01.006. Epub 2007 Apr 24. PMID 17459741
- [Background] Siev-Ner I, Gamus D, Lerner-Geva L, Achiron A. Reflexology treatment relieves symptoms of multiple sclerosis: a randomized controlled study. Mult Scler. 2003 Aug;9(4):356-61. doi: 10.1191/1352458503ms925oa. PMID 12926840
- [Background] Holt J, Lord J, Acharya U, White A, O'Neill N, Shaw S, Barton A. The effectiveness of foot reflexology in inducing ovulation: a sham-controlled randomized trial. Fertil Steril. 2009 Jun;91(6):2514-9. doi: 10.1016/j.fertnstert.2008.04.016. Epub 2008 Jun 20. PMID 18565520
- [Background] Sudmeier I, Bodner G, Egger I, Mur E, Ulmer H, Herold M. [Changes of renal blood flow during organ-associated foot reflexology measured by color Doppler sonography]. Forsch Komplementarmed. 1999 Jun;6(3):129-34. doi: 10.1159/000021238. German. PMID 10460981
- [Background] Hughes CM, Krirsnakriengkrai S, Kumar S, McDonough SM. The effect of reflexology on the autonomic nervous system in healthy adults: a feasibility study. Altern Ther Health Med. 2011 May-Jun;17(3):32-7. PMID 22164810
- [Background] Sliz D, Smith A, Wiebking C, Northoff G, Hayley S. Neural correlates of a single-session massage treatment. Brain Imaging Behav. 2012 Mar;6(1):77-87. doi: 10.1007/s11682-011-9146-z. PMID 22261925
- [Background] McCullough JE, Liddle SD, Sinclair M, Close C, Hughes CM. The physiological and biochemical outcomes associated with a reflexology treatment: a systematic review. Evid Based Complement Alternat Med. 2014;2014:502123. doi: 10.1155/2014/502123. Epub 2014 May 5. PMID 24883067